CLINICAL TRIAL: NCT00001502
Title: Pediatric Phase I Trial of RMP-7 and Carboplatin in Brain Tumors
Brief Title: A Pediatric Phase I Trial of RMP-7 and Carboplatin in Brain Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 960068; 96-C-0068
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2000-02

CONDITIONS: Brain Neoplasms; Glioma; Medulloblastoma
Keywords: Blood-Brain Barrier; Bradykinin; Children; Glioma; Medulloblastoma
MeSH Terms: conditions — Brain Neoplasms; Glioma; Medulloblastoma | interventions — RMP 7; Carboplatin

INTERVENTIONS:
Drug: RMP-7 and carboplatin

SUMMARY:
The presence of a highly selective blood-brain barrier (BBB) at the level of the brain capillary endothelium prevents chemotherapeutic agents from attaining therapeutic concentrations at the target site. RMP-7 is a synthetic bradykinin analog which specifically binds to B2 receptors expressed on the brain capillary endothelial cells and preferentially increases capillary permeability within CNS tumors. Carboplatin is an anticancer agent with preclinical and clinical antitumor activity against a variety of brain tumors. A pediatric phase I trial of the combination of RMP-7 and carboplatin will be conducted to determine the maximum tolerated dose of RMP-7 in children with refractory brain tumors.

DETAILED DESCRIPTION:
The presence of a highly selective blood-brain barrier (BBB) at the level of the brain capillary endothelium prevents chemotherapeutic agents from attaining therapeutic concentrations at the target site. RMP-7 is a synthetic bradykinin analog which specifically binds to B2 receptors expressed on the brain capillary endothelial cells and preferentially increases capillary permeability within CNS tumors. Carboplatin is an anticancer agent with preclinical and clinical antitumor activity against a variety of brain tumors. A pediatric phase I trial of the combination of RMP-7 and carboplatin will be conducted to determine the maximum tolerated dose of RMP-7 in children with refractory brain tumors.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

Histologically confirmed brain tumor including but not limited to the following: Anaplastic astrocytoma, Glioblastoma multiforme, Low-grade glioma, Ependymoma, Medulloblastoma, Pineal tumors, Chiasmal glioma, Craniopharyngioma, Brain stem glioma (requirement for histologic diagnosis may be waived).

Disease refractory to standard therapy or no standard chemotherapy exists and ineligible for potential curative surgery or radiotherapy.

Measurable or evaluable disease on radiographic studies with evidence of progression on prior chemotherapy or radiotherapy or persistent disease after surgery.

PRIOR/CURRENT THERAPY:

See Disease Characteristics

At least 6 months since carboplatin.

At least 3 weeks since myelosuppressive therapy.

Patients who received stem cell or bone marrow rescue after nitrosourea therapy are eligible after 3 weeks if they have recovered from hematologic toxicities of their prior therapy.

Concurrent steroids allowed if dose stable for at least 2 weeks prior to entry.

Recovered from toxic effects of any prior therapy.

PATIENT CHARACTERISTICS:

Age: 21 and under.

Performance status: ECOG 0-2.

Life expectancy: At least 8 weeks.

HEMATOLOGIC:

Absolute granulocyte count greater than 1,500/mm(3).

Platelet count greater than 100,000/mm(3) (at least 75,000/mm(3) in patients with prior bone marrow transplantation or craniospinal irradiation).

Hemoglobin greater than 8.0 g/dL.

HEPATIC:

Bilirubin no greater than 2 times normal.

ALT no greater than 2 times normal.

RENAL:

Creatinine within normal limits for age as follows:

Age (in years) -- Creatinine (in mg/dL):

Younger than 5 -- no greater than 1.2;

5-10 -- no greater than 1.5;

10-15 -- no greater than 1.8;

Older than 15 -- no greater than 2.4.

OTHER:

No significant systemic illness.

No pregnant or nursing women.

Negative pregnancy test required of fertile women.

Effective contraception required of fertile patients.

Durable power of attorney required of all patients 18-21 years of age.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30
Dates: Start 1996-04; Study Completion 2000-03

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Clements JA. The human kallikrein gene family: a diversity of expression and function. Mol Cell Endocrinol. 1994 Feb;99(1):C1-6. doi: 10.1016/0303-7207(94)90138-4. No abstract available. PMID 8187947
- [Background] Straub JA, Akiyama A, Parmar P. In vitro plasma metabolism of RMP-7. Pharm Res. 1994 Nov;11(11):1673-6. doi: 10.1023/a:1018986510570. No abstract available. PMID 7870689
- [Background] Inamura T, Nomura T, Bartus RT, Black KL. Intracarotid infusion of RMP-7, a bradykinin analog: a method for selective drug delivery to brain tumors. J Neurosurg. 1994 Nov;81(5):752-8. doi: 10.3171/jns.1994.81.5.0752. PMID 7931623